CLINICAL TRIAL: NCT06327490
Title: A Pilot Study Evaluating the Feasibility and Compliance of Manual Lymphatic Drainage Comparing Indocyanine-Green (ICG) Guided vs. Traditional Guided in Patients Undergoing Axillary Node Dissection for the Treatment of Breast Cancer
Brief Title: A Study Evaluating the Feasibility and Compliance of Manual Lymphatic Drainage Comparing Indocyanine-Green (ICG) Guided vs. Traditional Guided in Patients Undergoing Axillary Node Dissection for the Treatment of Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UF-BRE-012; IRB202400626 (Other: University of Florida); OCR44989 (Other: University of Florida)
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: breast cancer-related lymphedema; ICG-Lymphography Guided Manual Lymphatic Drainage; limb volume changes
MeSH Terms: conditions — Breast Neoplasms; Breast Cancer Lymphedema | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ICG-guided manual lymphatic drainage (Experimental)
  Interventions: Procedure: ICG-guided manual lymphatic drainage; Drug: Indocyanine green
- Traditional manual lymphatic drainage (Active Comparator)
  Interventions: Procedure: Traditional manual lymphatic drainage

INTERVENTIONS:
Procedure: ICG-guided manual lymphatic drainage — Participants will perform manual lymphatic drainage on their affected arm using ICG lymphography images of the lymphatic pathway in their affected arm as guidance once daily for 2 years post-surgery.
  Arms: ICG-guided manual lymphatic drainage
Procedure: Traditional manual lymphatic drainage — Participants will perform manual lymphatic drainage on their affected arm using traditional technique once daily for 2 years post-surgery.
  Arms: Traditional manual lymphatic drainage
Drug: Indocyanine green — All participants will be injected with indocyanine green for lymphatic mapping of the affected upper extremity, however this mapping will only be used to guide manual lymphatic drainage for participants on the ICG-guided manual lymphatic drainage arm.
  Arms: ICG-guided manual lymphatic drainage

SUMMARY:
Breast cancer is estimated to affect approximately 300,000 women in the US in 2023. Studies demonstrate that 1 in 5 will develop breast cancer related lymphedema secondary to the treatments that they receive. BCRL at this time has no cure, however early detection can prevent the progression to late stage BCRL. At this time a technique of arm massage, manual lymphatic drainage (MLD), is used for treatment. This study investigates a new method of MLD, which is guided by the individual patients' lymphatic anatomy through use of ICG-lymphography.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age
* Patients undergoing axillary lymph node dissection with or without lymphatic reconstruction at diagnosis
* Patients must have ICG lymphatic mapping performed prior to axillary lymph node dissection
* A clinical diagnosis consistent with stage Tis-T4N0-3M0 breast cancer.
* ECOG Performance Status of 0-1
* Subjects must not have more than one active malignancy at the time of enrollment (Subjects with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen [as determined by the treating physician and approved by the PI] may be included).
* Written informed consent obtained from the subject and the subject agrees to comply with all the study-related procedures.
* Subjects of childbearing potential (SOCBP) must have a negative pregnancy test prior to enrollment and be using an adequate method of contraception to avoid pregnancy throughout study participation to minimize the risk of pregnancy. Prior to study enrollment, subjects of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy.
* Patients must undergo a baseline physical therapy evaluation prior to axillary lymph node dissection.
* Patients who have received neoadjuvant chemotherapy are required to see physical therapy for lymphedema assessment following completion of chemotherapy prior to surgery.

Exclusion Criteria:

* Patients with history of ipsilateral breast cancer (invasive or ductal carcinoma in situ (DCIS))
* Patients with history of prior ipsilateral axillary surgery, such as excisional biopsy of lymph nodes or treatment of benign axillary disease processes such as hidradenitis
* Patients with history of or concurrent diagnosis of contralateral breast cancer (bilateral breast cancer)
* Patients with planned contralateral axillary surgery or history of contralateral axillary surgery
* Patients with a history, or concurrent, malignancy of the ipsilateral upper extremity- i.e. skin cancer
* Patients with history of lymphedema or lymphatic dysmotility of the ipsilateral or contralateral arm or are found to have lymphatic dysfunction at their pre-operative visit
* Patients with history of upper extremity blood clot, lymphangitis/cellulitis
* Patients with history of congestive heart failure or significant cardiac disease (such as New York Heart Association Class III or greater cardiac disease) including pacemakers incompatible for bioimpedance
* Patients with history of allergy to ICG or Iodine/Shellfish
* Patients with evidence of liver dysfunction including diagnosis of end stage liver disease
* Patients with less than 10 lymph nodes removed if no neoadjuvant chemotherapy (NAC) received, or less than 8 lymph nodes if NAC received. These node counts include nodes harvested as part of sentinel lymph node biopsy
* There is a lack of description of intraoperative findings during axillary lymph node dissection, such as the absence of notes on anatomy and procedure.
* Patients who are confirmed to be pregnant or breastfeeding.
* History of any other disease, metabolic dysfunction, clinical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of protocol therapy or that might affect the interpretation of the results of the study or that puts the subject at high risk for treatment complications, in the opinion of the treating physician.
* Prisoners or subjects who are involuntarily incarcerated, or subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Subject compliance | 2 years
  Determine subject compliance rate with daily manual lymphatic drainage regimen. A subject is considered to be compliant if they perform manual lymphatic drainage at least 3 days/week.

SECONDARY OUTCOMES:
Relative volume change | 2 years
  Determine if patients undergoing ICG-guided MLD as compared to patients undergoing traditional MLD demonstrate reduced relative volume changes of the affected limb. The volume of the affected limb will be measured by circumferential limb measurements. These limb measurements will then be calculated into volume using conic geometry.
Bioimpedance | 2 years
  Determine if patients undergoing ICG-guided MLD as compared to patients undergoing traditional MLD demonstrate lower rates of increased bioimpedance. Bioimpedance will be measured using both the sozo and in-body device methods.
Breast cancer related lymphedema symptoms | 2 years
  Determine if patients undergoing ICG-guided MLD as compared to patients undergoing traditional MLD demonstrate lower rates of breast cancer related lymphedema symptoms. Breast cancer related lymphedema symptoms will be assessed by the Lymphedema Life Impact Scale questionnaire.
Incidence of progression to late stage breast cancer related lymphedema | 2 years
  Compare the incidence of progression to late stage breast cancer related lymphedema in both arms
Health-related quality of life | 2 years
  Compare health-related quality of life, as measured by the Lymphedema Life Impact Scale questionnaire, in both arms.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Spiguel, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States